CLINICAL TRIAL: NCT01677650
Title: The Influence of Pharmacogenetics on Methadone Dose, Safety, and Outcomes After Spine Fusion
Brief Title: Pharmacogenomics of Methadone in Spine Fusion Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator moved to new institution
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dhanesh Gupta, Associate Professor of Anesthesiology & Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00064915
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Scoliosis; Kyphosis
Keywords: Spinal Fusion; Opioid Analgesia
MeSH Terms: conditions — Scoliosis; Kyphosis | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Methadone 0.5 mg/kg (Active Comparator): Methadone 0.5 mg/kg
  Interventions: Drug: Methadone
- Methadone 0.4 mg/kg (Experimental): Methadone 0.4 mg/kg
  Interventions: Drug: Methadone
- Methadone 0.3 mg/kg (Active Comparator): Methadone 0.3 mg/kg
  Interventions: Drug: Methadone
- Methadone 0.2 mg/kg (Active Comparator): Methadone 0.2 mg/kg
  Interventions: Drug: Methadone
- Methadone 0.15 mg/kg (Active Comparator): Methadone 0.15 mg/kg
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Methadone IV Pre-Induction of Anesthesia 0.15 to 0.5 mg/kg
  Other Names: Dolophine

SUMMARY:
The overall objective is to develop a patient oriented research program to efficiently evaluate the effects of pharmacogenetic variants on the dose-response relationships and safety of opioids and non-opioid analgesics. If an opioid regimen can be created that produces excellent opioid analgesia with minimal toxicity related to supratherapeutic opioid concentrations (i.e., ventilatory depression), other non-opioid analgesics (i.e., gabapentin/pregabalin, ketamine, lidocaine, cyclooxygenase inhibitors, etc.) that may decrease preoperative opioid requirements can be more efficiently and safely evaluated. These interventions may limit the opioid related toxicities related to effect site concentrations that are below those required when opioids are the predominant analgesic, such as opioid related ileus. Methadone's slow elimination clearance and limited pharmacokinetic drug-drug interactions make it an attractive perioperative opioid. The first step towards personalized opioid analgesia is to determine the effect of common pharmacogenetic variants that affect either methadone metabolism (CYP2B6) or opioid elimination.

DETAILED DESCRIPTION:
This study is being done to find the optimal dose of methadone (a long acting pain medication) that decreases the amount of pain that people have after spine surgery. Five different doses of methadone will be compared to each other, while keeping the remainder of the anesthetic routine for surgery. The investigators will determine the analgesic dose-response of methadone. The investigators will also determine the effect of methadone on the incidence of opioid related side effects, the quality of outcome of recovery, and the change in the 3-month opioid use.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II, and III
* male and non-pregnant female
* English-speaking
* undergoing elective < 3 vertebral level lumbar spine fusion (with and without interbody fusion)

Exclusion Criteria:

* Use of more than the equivalent of 20 mg of IV morphine/24 hr in the past 2 weeks
* history of substance abuse at any time in the past
* known QT prolongation
* Non-elective operations (i.e., cancer or trauma)
* severe hepatic impairment (serum albumin <3.0 g/dL, history of liver disease)
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Time until initial request for postoperative analgesic. | 60 minutes after extubation, 24, 48, and 72 hours after methadone administration

SECONDARY OUTCOMES:
The determination of minimum effective analgesic concentration of methadone. | 60 minutes after extubation, 24, 48, and 72 hours after methadone administration
Postoperative pain at rest and with movement (numerical rating scale, NRS) | 60 minutes after extubation, 24, 48, and 72 hours after methadone administration
The number of occurrences of ventilatory depression during each evaluation interval | 60 minutes after extubation, 24, 48, and 72 hours after methadone administration
Nausea and vomiting: number of rescue antiemetic doses and episodes of emesis | 60 minutes after extubation, 24, 48, and 72 hours after methadone administration
Level of sedation (modified Observer's Assessment of Alertness and Sedation Scale, modified OAA/S scale) | 60 minutes after extubation, 24, 48, and 72 hours after methadone administration
Occurence of pruritis | 60 minutes after extubation, 24, 48, and 72 hours after methadone administration
Algometry to assess pain tolerance | Pre-operatively, 60 minutes after extubation, 24, 48, and 72 hours after methadone administration
Degree of bother associated with opioid-related adverse effects: Opioid-related Symptom Distress Scale (OR-SDS) | 24, 48, and 72 hours after methadone administration
Quality of Recovery: Quality of Recovery-40 score | 24, 48, and 72 hours after methadone administration
Patient analgesic satisfaction | 24, 48, and 72 hours after methadone administration
Assessment of back condition pre and post-operatively | Pre-operatively, 6 weeks and 3 months post-operatively
Effects of common opioid related metabolic pathway polymorphisms on methadone's dose response relationships for analgesia and side effects | Preoperatively
  CYP2B6 Polymorphism effect on
  1. Time to first request for analgesia
  2. Secondary outcomes
Pupillometry for assessment of sedation | Pre-operatively, 60 minutes after extubation, 24, 48, and 72 hours after methadone administration

CONTACTS AND LOCATIONS:
Overall Officials: Dhanesh K. Gupta, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Rajaee SS, Bae HW, Kanim LE, Delamarter RB. Spinal fusion in the United States: analysis of trends from 1998 to 2008. Spine (Phila Pa 1976). 2012 Jan 1;37(1):67-76. doi: 10.1097/BRS.0b013e31820cccfb. PMID 21311399
- [Background] Jadad AR, Browman GP. The WHO analgesic ladder for cancer pain management. Stepping up the quality of its evaluation. JAMA. 1995 Dec 20;274(23):1870-3. PMID 7500538
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Upton RN, Semple TJ, Macintyre PE. Pharmacokinetic optimisation of opioid treatment in acute pain therapy. Clin Pharmacokinet. 1997 Sep;33(3):225-44. doi: 10.2165/00003088-199733030-00005. PMID 9314613
- [Background] Taylor S, Kirton OC, Staff I, Kozol RA. Postoperative day one: a high risk period for respiratory events. Am J Surg. 2005 Nov;190(5):752-6. doi: 10.1016/j.amjsurg.2005.07.015. PMID 16226953
- [Background] Taylor S, Voytovich AE, Kozol RA. Has the pendulum swung too far in postoperative pain control? Am J Surg. 2003 Nov;186(5):472-5. doi: 10.1016/j.amjsurg.2003.07.021. PMID 14599609
- [Background] Liu N, Kuhlman G, Dalibon N, Moutafis M, Levron JC, Fischler M. A randomized, double-blinded comparison of intrathecal morphine, sufentanil and their combination versus IV morphine patient-controlled analgesia for postthoracotomy pain. Anesth Analg. 2001 Jan;92(1):31-6. doi: 10.1097/00000539-200101000-00007. PMID 11133596
- [Background] Joris J, Kaba A, Lamy M. Transition between anesthesia and post-operative analgesia: relevance of intra-operative administration of analgesics. Acta Anaesthesiol Belg. 2001;52(3):271-9. PMID 11732383
- [Background] Carroll IR, Angst MS, Clark JD. Management of perioperative pain in patients chronically consuming opioids. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):576-91. doi: 10.1016/j.rapm.2004.06.009. PMID 15635517
- [Background] Yaksh TL, Hua XY, Kalcheva I, Nozaki-Taguchi N, Marsala M. The spinal biology in humans and animals of pain states generated by persistent small afferent input. Proc Natl Acad Sci U S A. 1999 Jul 6;96(14):7680-6. doi: 10.1073/pnas.96.14.7680. PMID 10393880
- [Background] Parker RK, Holtmann B, White PF. Effects of a nighttime opioid infusion with PCA therapy on patient comfort and analgesic requirements after abdominal hysterectomy. Anesthesiology. 1992 Mar;76(3):362-7. doi: 10.1097/00000542-199203000-00007. PMID 1539846
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Chui PT, Gin T. A double-blind randomised trial comparing postoperative analgesia after perioperative loading doses of methadone or morphine. Anaesth Intensive Care. 1992 Feb;20(1):46-51. doi: 10.1177/0310057X9202000109. PMID 1609941
- [Background] van Dorp EL, Kest B, Kowalczyk WJ, Morariu AM, Waxman AR, Arout CA, Dahan A, Sarton EY. Morphine-6beta-glucuronide rapidly increases pain sensitivity independently of opioid receptor activity in mice and humans. Anesthesiology. 2009 Jun;110(6):1356-63. doi: 10.1097/ALN.0b013e3181a105de. PMID 19461298
- [Background] Egan TD, Huizinga B, Gupta SK, Jaarsma RL, Sperry RJ, Yee JB, Muir KT. Remifentanil pharmacokinetics in obese versus lean patients. Anesthesiology. 1998 Sep;89(3):562-73. doi: 10.1097/00000542-199809000-00004. PMID 9743391
- [Background] Lemmens HJ, Brodsky JB, Bernstein DP. Estimating ideal body weight--a new formula. Obes Surg. 2005 Aug;15(7):1082-3. doi: 10.1381/0960892054621350. PMID 16105412
- [Background] Bowdle TA, Even A, Shen DD, Swardstrom M. Methadone for the induction of anesthesia: plasma histamine concentration, arterial blood pressure, and heart rate. Anesth Analg. 2004 Jun;98(6):1692-1697. doi: 10.1213/01.ANE.0000114085.20751.20. PMID 15155330
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Apfelbaum JL, Gan TJ, Zhao S, Hanna DB, Chen C. Reliability and validity of the perioperative opioid-related symptom distress scale. Anesth Analg. 2004 Sep;99(3):699-709. doi: 10.1213/01.ANE.0000133143.60584.38. PMID 15333398
- [Background] Myles PS, Hunt JO, Fletcher H. Measuring health status (quality of recovery?) after anesthesia and surgery. Anesth Analg. 2001 Jan;92(1):281. doi: 10.1097/00000539-200101000-00062. No abstract available. PMID 11133650
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Chou WY, Wang CH, Liu PH, Liu CC, Tseng CC, Jawan B. Human opioid receptor A118G polymorphism affects intravenous patient-controlled analgesia morphine consumption after total abdominal hysterectomy. Anesthesiology. 2006 Aug;105(2):334-7. doi: 10.1097/00000542-200608000-00016. PMID 16871067
- [Background] Romberg RR, Olofsen E, Bijl H, Taschner PE, Teppema LJ, Sarton EY, van Kleef JW, Dahan A. Polymorphism of mu-opioid receptor gene (OPRM1:c.118A>G) does not protect against opioid-induced respiratory depression despite reduced analgesic response. Anesthesiology. 2005 Mar;102(3):522-30. doi: 10.1097/00000542-200503000-00008. PMID 15731588